CLINICAL TRIAL: NCT05744271
Title: Evaluation of FES+VFBT With Individuals With Lived Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-5868
Record Dates: First submitted 2023-01-18; First posted 2023-02-24 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injuries; Stroke
Keywords: Balance; Functional Electrical Stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Stroke

STUDY DESIGN:
Intervention Model Description: A single-subject design will be used, allowing each participant to be his/her own control. Repeated assessments will be taken over three periods: a baseline (i.e. no intervention), intervention, and follow-up.
Masking Description: Performance on clinical measures will be evaluated by a physical therapist who is blind to the study purpose, design, and intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FES+VFBT (Experimental): Functional electrical stimulation combined with visual feedback balance training
  Interventions: Device: FES+VFBT

INTERVENTIONS:
Device: FES+VFBT — Standing balance training with the FES+VFBT system will occur 3x/week for six weeks (i.e. 18 sessions). Electrodes will be placed on the participants' plantarflexors and dorsiflexors bilaterally and FES will be administered using the device, MyndSearch, during the balance training exercises. Each session will last one hour, including 15 min to identify motor thresholds and maximum tolerable stimulation levels, 5 min to don/doff the safety harness, 5 min to calibrate the FES+VFBT exercises, 20 min to complete the FES+VFBT exercises, and 10-15 min to take rest breaks between exercises as needed.

SUMMARY:
Falls are an "emerging public health crisis" that cost the Canadian health care system billions of dollars each year. Moreover falls have a significant, detrimental impact on the lives of those who fall. In addition to physical injury and hospital admission, individuals may experience a post-fall syndrome characterized by dependence, depression, and reduced mobility and participation. Individuals living with the effects of neurological disease or injury are at a particularly high risk of falling. For example, 69-78% of individuals with spinal cord injury or disease (SCI/D) and 73% of individuals post-stroke fall at least once per year. Despite this high fall risk, evidence-based initiatives to prevent falls among those with SCI/D or stroke are lacking in neurorehabilitation. Furthermore, little time is dedicated to improving balance during inpatient neurorehabilitation. For example, ambulatory inpatients with SCI/D spend, on average, a mere 2.0±2.0 hours on balance training over the course of their entire inpatient stay. Our team is developing effective solutions to the "high-volume, high-risk and high-cost challenge" of falls. Our long-term objective is to develop an intervention that improves balance in a clinically meaningful and feasible way, facilitating the recovery of safe upright mobility and addressing the current health crisis of falls in individuals living with neurological disease or injury. The intervention will be developed with a focus on neurological populations, as these patient groups have a critical need for balance training; however, the intervention will be transferrable to other populations at risk of falls, such as older able-bodied adults.

A probable solution to the gap in balance interventions is functional electrical stimulation (FES), whereby an electrical current is applied to peripheral nerves to facilitate muscle contractions. By applying the appropriate amount of electrical stimulation at the appropriate time during movement execution, the central nervous system can be re-educated, facilitating motor and functional improvements. The investigators developed a closed-loop FES system whose controller mimics the physiological control system. By combining this system with visual feedback balance training (VFBT), the investigators developed a prototype system of FES and VFBT (FES+VFBT). This intervention involves standing on a force plate with one's centre of pressure (COP) presented on a monitor. As the user moves his/her COP in response to a game, FES is delivered to the plantarflexor and dorsiflexor muscles through the device, MyndSearch.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with a non-progressive, motor incomplete SCI/D (i.e. American Spinal Injury Association Impairment Scale (AIS) C or D) or a middle cerebral artery (MCA) stroke
2. chronic stage of recovery (i.e. >1 year post-SCI/D or stroke), when natural recovery has plateaued
3. ≥18 years old
4. able to stand independently for 60 seconds
5. moderate level of trunk control as evidenced by the ability to reach forward >2 inches in standing (i.e. score of 1-3 on the Berg Balance Scale Reaching Forward task);
6. free of any other condition besides SCI/D or stroke that significantly affects walking or balance (e.g., no vestibular disorder, significant vision loss)
7. able to understand spoken English

Exclusion Criteria:

1. a prior lower extremity fragility fracture
2. an injection of botulinum toxin to leg muscles in the past two weeks or injection planned during treatment period
3. peripheral nerve damage in the legs
4. contraindications for FES (i.e. implanted electronic device, active cancer or radiation in past six months, uncontrolled epilepsy, skin rash/wound at an electrode site, pregnancy, active deep vein thrombosis)31
5. contraindications for TMS (i.e. history of epilepsy and/or seizures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Change in Berg Balance Scale score | Baseline, after three weeks of the intervention, immediately after the intervention, 6-week follow-up after the intervention, 12-week follow-up after the intervention
  Scores range from 0-56, higher score equals greater balance
Change in Activities-specific Balance Confidence Scale score | Baseline, after three weeks of the intervention, immediately after the intervention, 6-week follow-up after the intervention, 12-week follow-up after the intervention
  Scores range from 0-100%, higher score equals greater confidence in balance
Change in strength of the trunk and lower extremity | Baseline, after three weeks of the intervention, immediately after the intervention, 6-week follow-up after the intervention, 12-week follow-up after the intervention
  The force, measured in lbs or kg, of eight lower extremity muscle groups (i.e. hip extensors, hip flexors, hip abductors, hip adductors, knee extensors, knee flexors, ankle plantarflexors and ankle dorsiflexors) will be measured using a hand-held dynamometer. Scores range from 0-40, higher score equals greater strength.
Change in static standing balance | Baseline, after three weeks of the intervention, immediately after the intervention, 6-week follow-up after the intervention, 12-week follow-up after the intervention
  Will be assessed by measuring postural sway during quiet standing on the force sensing mat for 60 seconds under two conditions presented in a random order: eyes open and eyes closed. The amount of body sway, such as COP amplitude and speed, will be quantified to examine the change of static balance as well as reliance on the visual information.
Change in dynamic standing balance | Baseline, after three weeks of the intervention, immediately after the intervention, 6-week follow-up after the intervention, 12-week follow-up after the intervention
  Will be assessed by asking participants to lean as far as possible in the forward, backward and sideways directions while standing on the force sensing mat (i.e. limits of stability test). The maximum centre of pressure (COP) amplitude in the anterior, posterior and mediolateral directions will be recorded. The change of COP amplitude will be assessed. Electromyography will be recorded in the major leg muscles. The change in co-contraction and muscle synergy will be investigated to quantify the change in muscle activation pattern by the intervention.
Questionnaire on the participants' perspectives of the FES+VFBT intervention | Immediately after the intervention
Semi-structured interview on the participants' perspectives of the FES+VFBT intervention | Immediately after the intervention

SECONDARY OUTCOMES:
Change in cutaneous pressure sensation | Baseline, after three weeks of the intervention, immediately after the intervention, 6-week follow-up after the intervention, 12-week follow-up after the intervention
  Monofilaments of six different thicknesses will be applied in order of descending thickness. Each monofilament will be applied six times with the participant's eyes closed. Participants will indicate when they can feel pressure being applied. Total score is the number of correct responses (maximum score of 72: 6 monofilaments x 6 applications x 2 toes).Scores range from 0-72, greater score equals greater cutaneous pressure sensation.
Change in correct proprioception responses of the first metatarso-phalangeal and ankle joints | Baseline, after three weeks of the intervention, immediately after the intervention, 6-week follow-up after the intervention, 12-week follow-up after the intervention
  With participants' eyes closed, the therapist will slowly move each joint through 10 degrees of range of motion in either the extension/plantarflexion or flexion/dorsiflexion directions. Participants will indicate the direction of the movement (i.e. down or up, respectively). Six movements per joint will be performed, resulting in a total possible score of 24 (6 movements x 4 joints). Scores range from 0-24, greater score equals greater proprioception.
Change of corticospinal excitability | Baseline, after three weeks of the intervention, immediately after the intervention, 6-week follow-up after the intervention, 12-week follow-up after the intervention
  Motor evoked potential induced by transcranial magnetic stimulation (TMS) will be measured during sitting to examine the corticospinal excitability.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin E Musselman, PhD, Principal Investigator — KITE-Toronto Rehabilitation Institute, UHN
Locations (1):
- KITE-Toronto Rehabilitation Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No